CLINICAL TRIAL: NCT04630860
Title: A Randomized, Open-label, Multiple Ascending Dose Study in Patients With Advanced-stage Parkinson's Disease to Evaluate the Pharmacokinetics and Safety of LY03003 Following Intramuscular Injections
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of LY03003 in Patients With Advanced-stage PD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY03003/CT-CHN-106
Record Dates: First submitted 2020-11-05; First posted 2020-11-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; LY03003
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 56mg dose group (Experimental)
  Interventions: Drug: LY03003
- 84mg dose group (Experimental)
  Interventions: Drug: LY03003
- 112mg dose group (Experimental)
  Interventions: Drug: LY03003

INTERVENTIONS:
Drug: LY03003 — Rotigotine,extended-release microspheres

SUMMARY:
This study is to evaluate the pharmacokinetics and safety of LY03003 in patients with advanced-stage PD.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent must be given to the study and written informed consent must be voluntarily signed, good communication with the investigator and compliance with all requirements of the clinical trial (planned visits, laboratory tests and other test procedures);
2. During screening, subjects are 18-80 years old (including boundary value), regardless of gender;
3. Male subjects shall weigh no less than 50kg and female subjects shall weigh no less than 45kg. Body mass index within the range of 19~30kg/m2 (including critical value);
4. Meet the diagnostic criteria of MDS for primary Parkinson's disease with sick time more than 3 years. The diagnosis is based on the main symptoms-motor retardation, plus at least one of the following symptoms: quiescence tremor, myotonia, and no other known or suspected causes of Parkinson's disease;
5. In the "on" state, subjects' HOehn-YahR rating is from level 2 to level 3;
6. A concise Mental State Scale (MMSE) score ≥25;
7. A steady dose of Levodopa (either monotherapy or in combination with benserazide/carbidopa/carbidopa) shall be administered at least 2 times a day for a minimum of 28 days prior to baseline;
8. if you are accept anticholinergic drugs (such as benzalkonium tropic, benzene hai suo, diethyl promethazine, its organism and than pp board), monoamine oxidase B (MAO B) inhibitors (e.g., company to gillan, LeiSha gillan) and/or N - methyl - d - aspartate (NMDA) antagonist (such as amantadine) treatment, must be accepted before baseline at least 28 days, stable doses and during the study period to maintain the therapeutic dose;
9. Women of childbearing age (those who do not meet any of the following conditions: menstrual stop ≥ 12 months; Or had undergone hysterectomy or bilateral oophorectomy; (or with medically confirmed ovarian failure) or male subjects agree to use reliable contraceptives (oral contraceptives, condom use, abstinence, etc.) throughout the study period (screening visits until the end of the study), and pregnancy tests for women of childbearing age are negative at screening and baseline.

Exclusion Criteria:

1. Patients with atypical Parkinson's disease caused by the use of drugs (such as methoxylopramine, flunarizine), hereditary metabolic diseases of the nervous system (such as Wilson's disease), encephalitis, cerebrovascular diseases or degenerative diseases (such as progressive supravuclear palsy);
2. The author had a history of epilepsy, or had a history of stroke or transient ischemic stroke within 1 year before the visit;
3. Dementia, active mental illness or hallucinations, major depression;
4. Those with a history of suicide attempts (including actual attempts, attempts interrupted or failed) or suicidal ideation in the past 6 months, defined as those who answered "yes" to question 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at the time of screening;
5. Patients with a history of narcolepsy;
6. There is impulse control disorder (ICD) evidence;
7. Uncontrolled or severe cardiovascular disease, including New York Heart Association (NYHA) class II or higher congestive heart failure, unstable angina, myocardial infarction, or the presence of arrhythmia requiring treatment during screening;
8. Patients with malignant tumors within 5 years before screening, except for cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, local prostate cancer after radical surgery, and intraductal carcinoma in situ after radical surgery;
9. History of pallidotomy, thalamic lesion, deep brain stimulation or fetal tissue transplantation;
10. received cabergoline or bromocriptine within 15 days before baseline, or received other dopamine agonists within 7 days before baseline;
11. Patients received any of the following drugs within 28 days before baseline: α-methyldopa, metoclopramide, flunarizine, reserpine, antipsychotics, monoamine oxidase A (MAO-A) inhibitors, methylphenidate, amphetamine, cloth, etc.;
12. Currently receiving treatment for central nervous system diseases (e.g., sedatives, hypnotics, antidepressants, anxiolytics), unless the dose is stable for at least 28 days before baseline, and the treatment dose is maintained during the study period;
13. Known history of intolerance/allergy to the following antiemetics: domperidone, trimethoxybenzamide, ondansetron, tropisetron, granisetron, and glycopyrrolate;
14. Screening or baseline, ECG examination QTc > 450 milliseconds (male) or > 460 milliseconds (female) or other abnormalities judged by the investigator have clinical significance;
15. History of orthostatic hypotension; or systolic blood pressure (SBP) decreased by ≥ 20 mmHg or diastolic blood pressure (DBP) decreased by ≥ 10 mmHg when changing from the decubitus position to the upright position for 1 or 3 minutes at screening or baseline; or systolic pressure < 105 mmHg at screening or baseline;
16. Clinically significant abnormal liver function, defined as total bilirubin > 1.5 times the upper limit of the reference range or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of the reference range;
17. Clinically significant renal dysfunction (serum creatinine > 2.0 mg/dL or > 177 umol/L]);
18. Any test result of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody is positive;
19. Smokers, alcoholics:

    A) Smoking is defined as: an average daily smoking of ≥ 5 cigarettes within 3 months before screening; B) Alcohol abuse is defined as: drinking more than 14 units of alcohol per week (1 unit = 350 mL of beer, or 45 mL of liquor, or 150 mL of wine) within 3 months before screening.
20. Pregnant or lactating women;
21. Allergic constitution (allergic to two or more drugs or food) or known to be allergic to rotigotine or rotigotine microsphere preparation ingredients;
22. Previous use of rotigotine-containing preparations can not tolerate or poor efficacy;
23. Participated in other drug clinical trials within 3 months before screening;
24. Other clinically significant medical conditions, mental conditions or laboratory abnormalities that may interfere with the ability of the subject to participate in this study as judged by the investigator;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Safety evaluation | From Titration Period to Day 50 of Dose Maintenance Period
  Blood pressure
Cmax ,ss | From Titration Period to Day 50 of Dose Maintenance Period
  Peak concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China